CLINICAL TRIAL: NCT06617624
Title: Magnetic Resonance Imaging Development for High Resolution Atrial Structural and Functional Characterization
Acronym: MRI-HiRA
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231076; 2023-A01951-44 (Other: ID-RCB)
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Patients with Atrial Fibrillation and Healthy Volunters
Keywords: Atrial fibrillation; MRI; Acquisition optimisation; Biomarkers
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group 1: patient with paroxysmal AF (Atrial Fibrillation) (no AF during exam): 20 patients able to complete the full standard experimental examination corresponding to paroxysmal AF group
  Interventions: Other: MRI Contrast
- Group 2: patient with persistent AF (Atrial Fibrillation): 20 patients able to complete the full standard experimental examination corresponding to persistent AF group
  Interventions: Other: MRI Contrast
- Group 3: patient with permanent AF (Atrial Fibrillation): 20 patients able to complete the full standard experimental examination corresponding to permanent AF group
  Interventions: Other: MRI Contrast
- Group 4: healthy volunteer: 60 age/sex BMI class matched healthy volunteers, able to complete the full standard experimental examination.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Healthy volunteer will have a non-injected cardiovascular MRI
  Groups: Group 4: healthy volunteer
Other: MRI Contrast — Patients will have the gadolinium injected cardiovascular MRI
  Groups: Group 1: patient with paroxysmal AF (Atrial Fibrillation) (no AF during exam); Group 2: patient with persistent AF (Atrial Fibrillation); Group 3: patient with permanent AF (Atrial Fibrillation)

SUMMARY:
The main objective is to optimize the MRI protocol for the assessment of the LA in addition to a basic CMR protocol in order to define the best compromise between acquisition time and image quality (contrast between the different tissues, spatial and temporal resolutions, etc.) sufficient for accurate measurement of morphological, structural and hemodynamic left atrial biomarkers.

DETAILED DESCRIPTION:
This Magnetic Resonance imaging study of the heart aims to acquire images and measures of:

1. Left atrial cine: compressed sensing cine imaging strategies will be tested for LA assessment by optimizing spatial and temporal resolution providing the best image quality relative to acceptable acquisition times. The whole heart should be covered during acquisition. Image quality and diagnosis of LA contraction preservation will be performed.
2. Myocardial tissue characterization including:

   1. 3D isotropic ECG-gated with respiratory navigation late gadolinium enhancement (LGE) sequence for high resolution imaging of myocardial injury and fibrosis.
   2. High resolution free-breathing T1/T2 mapping to quantify myocardial water content and measure native T1 relaxation and extracellular volume. 2D free breathing LGE will complement the protocol.
   3. Cardiac adipose tissue imaging will be performed using gated Dixon imaging. Pericardial adipose tissue (PAT) will be measured covering the whole heart including groove epicardial adipose tissue (EAT).
3. Flow measurements: test and optimize a 4D flow approach for the heart and aorta using compressed sensing and multi velocity encoding (VENC) encoding to insure high and precise multi-chamber velocity imaging(100, 150, 200, 250 cm/s). Two-chamber (including left appendage) in plane velocities will be compared between high resolution 2D and 4D. Of, note, such multi-VENC approach is mandatory for LA imaging because of the large heterogeneity of blood flow velocities within the LA during the cardiac cycle.
4. Technology validation: comparison of cardiac triggering using the beat sensor vs. surface ECG-gating will be tested as a means of improving patient experience and speed up MRI acquisition for subsequent population imaging.

This task will be performed at the Cardiovascular MRI Imaging Platform and Core Lab at the Pitié-Salpêtrière Hospital site by SU-ICAN & APHP (ICT), SU-LIB and SIEMENS partners with the goal to optimize, test and validate innovative approaches before wider application.

ELIGIBILITY:
Inclusion Criteria:

For all groups of AF patients:

* Over 18 years of age
* Participation to the MAESTRIA-AFNET 10 study
* Able to undergo an injected MRI examination
* Able to give consent
* Affiliated to French social security system

Specific inclusion criteria of AF patients (same as MAESTRIA-AFNET 10) Group 1: patients with paroxysmal AF (no AF during exam) clinically defined as AF episodes less than one week Group 2: patients with persistent AF, clinically defined as AF episodes longer than one week Group 3: patients with permanent AF, with no documented sinus rhythm or possibility to restore sinus rhythm by any means

For healthy volunteers (Group 4):

* Over 18 years of age (including 30 subjects < 60 years)
* Able to undergo an MRI examination
* Able to give consent
* Affiliated to French social security system

Exclusion Criteria:

For all groups

* Deprived of liberty or under legal protection (under guardianship or curatorship)
* Kidney disease with GFR <30 mL / min (because of the risks linked to the injection of DOTAREM ™ and iodine)
* Pregnant woman, breastfeeding, of childbearing age in the absence of effective contraception
* MRI contraindication (claustrophobia, patients with metallic foreign bodies)
* Participation to another interventional clinical trial (Jardé 1) For patients
* Patients with a history of renal disease (renal transplant, single kidney, renal cancer)
* Patients who have received a dose of contrast in the last 24 hours
* Patients who had a previous allergic or anaphylactic reaction to gadolinium For volunteers
* Subjects with known cardiovascular pathology or under cardiovascular treatment
* Subjects with cardiovascular history
* Subjects with cardiac rhythm or conduction disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 3 groups of patients and 1 control group: paroxysmal AF (atrial fibrillation) (no AF during exam), persistent AF, permanent AF and healthy controls.
  20 patients able to complete the full standard experimental examination corresponding to each AF group and 60 age/sex BMI class matched healthy volunteers, able to complete the full standard experimental examination.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of maximal Left Atrial (LA) longitudinal strain | 24 months
  Measurement of maximal Left Atrial (LA) longitudinal strain. Comparison between patients and healthy volunteers will allow to define normal values and thresholds for the given sequences.

SECONDARY OUTCOMES:
Various calibration settings against reference. | 24 months
  The metrics from the Linear regression and Bland and Altman analyses will be used to compare the various calibration settings against reference.
The correlation coefficients from the linear regressions | 24 months
  The correlation coefficients from the linear regressions will be estimated to assess the associations mentioned in the secondary objectives between the new biomarkers and the more established biomarkers.
The correlation coefficients from the linear regressions | 24 months
  The correlation coefficients from the linear regressions will be estimated to assess the associations mentioned in the secondary objectives between the new biomarkers and the more established biomarkers.Between LA imaging biomarkers and subcutaneous aging and pressure levels
ROC analysis | 24 months
  Metric of ROC analysis
The intra-operator coefficient of variation. | 24 months
  The intra-operator coefficient of variation.
The inter-operator coefficient of variation. | 24 months
  The inter-operator coefficient of variation.

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.